CLINICAL TRIAL: NCT02041312
Title: Serum Cholesterol and Gastric Neoplasm: Nested Case-control Study
Brief Title: Serum Cholesterol and Gastric Neoplasm
Acronym: SCGN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Yong Ahn, Professor, Asan Medical Center
Other Study IDs: AMC-1312; KCHUGRFG1312 (Other Grant/Funding Number: Korean J Helicobacter Up Gastrointest Res)
Record Dates: First submitted 2014-01-02; First posted 2014-01-22 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Gastric Cancer
Keywords: Cholesterol; Gastric cancer; Stage
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — endoscopic biopsy specimen of gastric mucosa surgically resected specimen of stomach
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gastric cancer: No intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention will be needed.

SUMMARY:
Investigators have a plan to conduct nested case-control study to investigate the association between serum cholesterol levels including TC, HDL-C, LDL-C, triglyceride (TG), apolipoproteins and gastric neoplasm. In addition, further analyses were performed to evaluate the possible role of the serum cholesterol as a predictor for the differentiation and prognosis of gastric neoplasm.

DETAILED DESCRIPTION:
Although its incidence has declined, gastric cancer remains one of the most common causes of cancer morbidity and mortality worldwide.Since the stage of gastric cancer at the time of detection correlates with prognosis, secondary prevention is important. Screening of asymptomatic individuals for gastric cancer has been shown to increase the detection of early gastric cancer (EGC), which has a 5-year overall survival (OS) rate exceeding 90%.

Gastric carcinogenesis is a multi-factorial process that includes environmental, socioeconomic, and lifestyle factors. Many of risk factors, including dietary factors, chronic atrophic gastritis, intestinal metaplasia, and H. pylori infection, alcohol consumption, and aspirin have been investigated. Although the specific correlation between serum cholesterol and gastric cancer is not fully understood, inverse relationships have been observed between serum total cholesterol (TC) levels and cancer, and recent analyses of randomized controlled trials showed significant inverse associations between high density lipoprotein cholesterol (HDL-C) and low density lipoprotein cholesterol (LDL-C) and the risk of incident cancers. Lower lipoprotein cholesterol in cancer patients may be due to the enhanced activity of the lipoprotein cholesterol receptor pathway and to the increased demand for cholesterol during tumor development and lymphatic spread. Some suggested that the preexisting tumor might have resulted in low serum cholesterol, which is called "preclinical cancer effect" or "unsuspected sickness". In another study, LDL-C has been reported to affect host immune system cells.

In our previous study, investigators found that serum HDL-C and LDL-C levels were associated with the risk, resectability, and prognosis of gastric cancer. There are several cohort studies reported that low serum cholesterol levels are associated with incident cancer, including gastric cancer. However, most studies regarding the serum cholesterol and gastric cancer investigated gastrectomized patients, and showed the association between low serum cholesterol levels and lymph node metastasis or submucosal invasion. Furthermore, there are only few studies evaluated the association between LDL-C of apolipoproteins and gastric cancer. Therefore investigators conducted nested case-control study to investigate the association between serum cholesterol levels including TC, HDL-C, LDL-C, triglyceride (TG), apolipoproteins and gastric neoplasm. In addition, further analyses were performed to evaluate the possible role of the serum cholesterol as a predictor for the differentiation and prognosis of gastric neoplasm.

ELIGIBILITY:
Inclusion Criteria:

* All subjects who visited the department of gastroenterology, surgery, or Healthcare Screening & Promotion Center at Asan Medical Center and diagnosed as gastric cancer

Exclusion Criteria:

* Subjects who has history about drug for cholesterol, diabetes, liver disease, and/or thyroid disease.
* Subjects who do not want to be enrolled this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects who visited the department of gastroenterology, surgery, or Healthcare Screening & Promotion Center at Asan Medical Center and diagnosed as gastric cancer
Sampling Method: Probability Sample
Enrollment: 1178 (Estimated)
Dates: Start 2014-02; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Cholesterol level in paitents with and withoutgastric neoplasm | up to 24 months
  Serum cholesterol levels including TC, HDL-C, LDL-C, triglyceride (TG), apolipoproteins will be checked and compared in paitents with and withoutgastric neoplasm.

SECONDARY OUTCOMES:
Degree of decresed serum cholesterol levels in paitents with gastric neoplasm | up to 24 months
  1. Degree of decresed serum cholesterol levels including TC, HDL-C, LDL-C, triglyceride (TG), apolipoproteins in patients with gastric neoplasm compare to the patients without gastric neoplasm.
  2. Degree of decresed serum cholesterol levels including TC, HDL-C, LDL-C, triglyceride (TG), apolipoproteins in patients with gastric neoplasm according to the stage of gastric neoplasm.

CONTACTS AND LOCATIONS:
Overall Officials: Hwoon-Yong Jung, M.D., PhD., Study Chair — Asan Medical Center
Locations (1):
- Department of Gastroenterology, University of Ulsan College of Medicine, Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No